CLINICAL TRIAL: NCT03027063
Title: Impact of Exercise on Mitigating the Cardio-toxic Effects of Adriamycin Among Women Newly Diagnosed With Breast Cancer Who Will be Treated With Anthracyclines
Brief Title: Impact of Exercise on Mitigating the Cardio-toxic Effects of Adriamycin Among Women Newly Diagnosed With Breast Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00110810
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer Female; Adriamycin Toxicity
Keywords: Speckle tracking echocardiography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10,000 steps (Experimental): For the "10,000 steps" group, participants will be asked to achieve a goal of 10,000 steps a day and to engage in 30 minutes of continuous exercise every day. Steps will be monitored with the under Armour fitness tracker which participants will receive.
  For motivation, messages will be sent to study participants in this group via the messaging center in the Under Armor application three times a week. The frequency of messaging will be increased for participants who fail to meet their goals for three consecutive days. Study participants will also receive a weekly call to assess for side effects and provide additional encouragement.
  Interventions: Behavioral: 10,000 steps
- Usual care (Active Comparator): This will be the usual care group. Participants will also receive a fitness tracker to enable monitoring of steps and will be given a flyer that references the ACC/AHA guidelines for exercise and physical activity for the general population. Participants will not receive text messages or phone calls.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: 10,000 steps — Participants will be asked to achieve 10,000 steps daily and to participate in 30 minutes of continuous exercise of their choosing. They will also receive text messages during the week and weekly motivational call
  Arms: 10,000 steps
Behavioral: Usual Care — Participants will receive the ACC/AHA exercise guidelines
  Arms: Usual care

SUMMARY:
This research is being done to determine whether exercise while receiving doxorubicin or Adriamycin chemotherapy for breast cancer can reduce the cardio-toxic effects of this treatment on the heart and improve other outcomes related to cancer such as tumor markers, nausea, fatigue and the ability to tolerate chemotherapy.

DETAILED DESCRIPTION:
This will be a pilot study that looks at the effect of exercise, while receiving anthracycline therapy, on mitigating the cardio toxic effects of anthracyclines as assessed by serial echocardiographic strain analysis.

Potential participants will be identified during chart review in advance of a routine clinic visit or during a routine clinic visit with a provider. Individuals will be approached by the provider or study team to determine willingness to learn more about a study for which they may be eligible. Discussions regarding study participation will take place privately and individuals will be provided with the Institutional Review Board (IRB) approved consent form.

In addition, potential participants may contact the study team directly. This contact may be in the form of telephone, email, etc. Initial discussions regarding study participation may take place by phone, email, etc., and individuals may be provided with the IRB approved consent form and other IRB reviewed and approved materials (e.g., Patient Handout), as applicable.

In all cases, as much time as is needed to consider study participation will be allowed to possible participants; resulting in multiple phone calls, visits, emails, or other communication, as necessary. For individuals who choose to take part, informed consent will happen as per the consent process.

Patients will be recruited from the Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Sibley Memorial Hospital and the community. The investigators anticipate that among roughly 60 subjects approached for enrollment, 30 will be part of the final study. Participants who agree to participate will be asked to provide written consent. Participants will be randomized by an online system to one of the following two groups in a 1:2 ratio. Group 1(Usual care group) will receive a fitness tracker and flyers that reference the American College of Cardiology/American Heart Association (ACC/AHA) guidelines for exercise and physical activity for the general population. In addition to fitness tracker and flyers, Group 2 (10,000 steps group) will receive additional messages and phone calls for motivation. This group of participants will also be asked to take part in 30 minutes of continuous exercise daily as part of their intervention.

For motivation, messages will be sent to study participants in group 2 via the messaging center in the Under Armour application three times a week. With the application, study participant will receive a phone alert and an email message to which they may respond if needed. The frequency of messaging will be increased for participants who fail to meet their goals for three consecutive days. In addition to the Under Armour application, participants will be provided with a log sheet for recording their daily steps, whether 30 minutes of continuous activity daily was completed and the type of the activity done for the 30 minutes. Group two study subjects will also receive a weekly call to assess for side effects and provide additional encouragement. Log sheets will be collected during oncology clinic visits and the aforementioned intervention will be continued for the duration of their chemotherapy treatment. Group 1 study participants will be assessed for side effects through a phone call every 4 weeks.

For the study, women will be given an Under Armour band that will monitor daily steps, amount of sleep and heart rate. Participants will be asked to download the Under Armour application to their mobile phones so the data from their bands can be synced with the application daily. For the intervention, study subjects will be asked to achieve a goal of 10,000 steps a day and to engage in 30 minutes of continuous exercise every day and this can be any form of exercise.

All patients who agree to participate will be invited to the Johns Hopkins Hospital medical campus where all the testing will be performed. The investigators expect to complete the study in 9 months.

Study participants who agree to participate will have the following assessments performed at baseline:

1. A Cardiopulmonary Exercise Stress Test done using the standard protocol and supervised by an exercise physiologist.
2. A 2D echocardiogram. The echocardiogram will include assessment of strain using speckle tracking and tissue Doppler and the determination of systolic ejection time. All patients routinely have an echocardiogram performed prior to the initiation of cardio-toxic chemotherapy such as doxorubicin (Adriamycin), trastuzumab (Herceptin) and pertuzumab (Perjeta), however, for the study, strain analysis will be performed off line on the images obtained during the clinically indicated baseline echocardiogram. Echocardiograms will be performed by experienced sonographers and on the same model echo machine to reduce variability.
3. Bone densitometry assessment via a Dual-energy X-ray absorptiometry to measure total and regional body composition in the frontal plane to determine bone, fat and fat-free mass. The Dual-energy X-ray absorptiometry scan takes about 8-10 minutes. The total radiation dose is approximately 1 millirem, which is very small.
4. Muscle strength will be measured using a hand grip tool.
5. Habitual activity levels will be assessed using the Rapid Assessment of Physical Activity questionnaire, which categorizes activity levels on a scale from 1-7 (sedentary to active).
6. Quality of life will be assessed with the Functional Assessment of Cancer Therapy-Breast survey
7. Fatigue level will be performed with the Multidimensional Fatigue Symptom Inventory-Short Form
8. All patients routinely have blood work collected, and as part of this research protocol, the investigators will also collect blood to determine baseline tumor markers ( high-sensitivity C-reactive protein, Insulin-like growth factor 1, interleukin -6, interleukin-1 and tumor necrosis factor alpha, leptin, adiponectin, estradiol, DNA extraction, lymphocyte telomere length) and cardiac biomarkers (high sensitivity troponin, troponin, pro-brain natriuretic peptide). The investigators will also collect and store blood in order to keep open the possibility of doing a more extensive study to look at any future genes that might be related to the phenotypes in this study (cancer, cardiomyopathy, exercise response, etc.).
9. Cardiac history will be obtained at recruitment, including clinical risk factors for heart disease (hypertension, diabetes and smoking history) and participants will be evaluated throughout the study for any cardiac symptoms especially those of Heart failure.

All of the above assessments will all be performed at baseline and repeated within 2 weeks of the women completing their anthracycline-based chemotherapy. The investigators will also track the clinical echocardiograms obtained at 12 months, but these results are not required for the study.

Other studies: Serum troponin levels will be checked with each cycle of chemotherapy. Height will be measured upon recruitment and weight and blood pressure will be measured at the time of each echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 years and older
* Women newly diagnosed with stage I to III breast cancer who will be receiving adjuvant or neoadjuvant doxorubicin-based chemotherapy
* Women who will be treated at the Johns Hopkins Hospital, Sibley Memorial Hospital or who will be treated by oncologists in the community as long as we will have access to treatment records.
* Women must be willing to receive follow up care either at Hopkins or with their local oncologist for at least 1 year.
* Patients who are receiving therapy with an anthracycline.
* Women who have a smart phone

Exclusion Criteria:

* Inability to exercise
* Presence of metastatic disease
* Advanced pulmonary disease as assessed by clinical symptoms of shortness of breath or known forced expiratory volume in 1 second < 1
* Any patients requiring oxygen at baseline
* The presence of known ischemic heart disease as defined by significant obstructive heart disease (stenosis > 70%) seen on coronary angiography or cardiac CT
* Abnormal baseline cardiac function defined as an ejection fraction of less than 55%
* The presence of more than mild valvular stenosis or regurgitation, prosthetic valves or pacemaker on their baseline echocardiogram
* Poor image quality on baseline echocardiogram or anatomic limitations that preclude the acquisition of good quality images such as recent mastectomy or surgery
* Patients who do not have a smart phone onto which the Under Armour application can be downloaded
* Patients who are unwilling to wear the Under Armour health band
* Pregnancy
* Previous anthracycline exposure
* Rhythms other than sinus rhythm
* Patients unwilling to come to the Johns Hopkins campus to have the required testing performed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Left ventricular dysfunction | Change from baseline to up to 14 weeks
  Development of left ventricular dysfunction, assessed by echocardiogram and defined as a decrease in global longitudinal strain between the baseline echocardiogram and the echocardiogram obtained post-treatment with an anthracycline.

SECONDARY OUTCOMES:
Cardiorespiratory fitness/peak oxygen consumption | Up to 14 weeks
  Cardiorespiratory fitness/peak oxygen consumption measured using a metabolic stress test
Dual-energy x-ray absorptiometry | Up to 14 weeks
  Dual-energy x-ray absorptiometry scan will be performed using standard procedures
Quality of life as assessed by the Functional Assessment of Cancer Therapy-Breast Survey | Up to 14 weeks
  Functional Assessment of Cancer Therapy-Breast survey will be administered upon completion of therapy to assess for change in quality of life. Each question on the questionnaire ranges from 0 to 4. The least score is 0 and the maximum is 148 points. Higher scores indicate a higher quality of life.
Physical Activity as assessed by the Rapid Assessment of Physical Activity Questionnaire | Up to 14 weeks
  Change in physical activity with the intervention will be assessed by the Rapid Assessment of Physical Activity questionnaire. This is scored from 1 to 7 with 7 being the most active.
Fatigue as assessed by the Multidimensional Fatigue Symptom Inventory-Short Form | Up to 14 weeks
  Multidimensional Fatigue Symptom Inventory-Short Form will be used to assess for change in fatigue. Scores for each question range from 0 to 4. The maximum total fatigue score is 72. The higher the score, the more fatigued one is.
Impact of motivational messages on increasing the amount of physical activity | Up to 14 weeks
  Analysis will be performed to assess the impact that receiving motivational text messages has on increasing the amount of physical activity performed/number of daily steps achieved.
Impact of telephone calls on increasing the amount of physical activity | Up to 14 weeks
  Analysis will be performed to assess the impact of weekly telephone calls on increasing the amount of physical activity/number of daily steps achieved
Impact of engaging in 30 minutes of exercise on increasing the amount of physical activity | Up to 14 weeks
  Analysis will be performed to assess the impact that engaging in 30 minutes of daily exercise has on increasing the amount of physical activity performed/number of daily steps achieved
Serum Troponin | Change from baseline to up to 14 weeks
  Difference in troponin levels in the the two groups post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Florido, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No